CLINICAL TRIAL: NCT01830114
Title: A Web App for Patients With Alcohol and Drug Use Problems in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Behavior Therapy Associates, LLP (Industry)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CheckupAndChoicesPilot; 1R43AA022024-01 (NIH)
Record Dates: First submitted 2013-04-08; First posted 2013-04-12 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Alcohol Abuse; Drug Abuse
Keywords: alcohol abuse; drug abuse; hazardous alcohol use; hazardous drug use
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Web app evaluation group (Experimental)
  Interventions: Behavioral: Web app

INTERVENTIONS:
Behavioral: Web app — The Checkup and Choices web application

SUMMARY:
The objective of this pilot study is to evaluate the feasibility and technical merit of a web application for patients in primary care called Check-up and Choices (CC).

DETAILED DESCRIPTION:
The overall objective of this project is to develop, evaluate, and disseminate a web application called Check-up and Choices (CC). CC will be developed for use in primary care. It would tightly integrate screening for heavy drinking and drug use, a brief motivational intervention for hazardous or heavy drinkers, a moderation training protocol for less dependent problem drinkers, and an abstinence-oriented protocol for more dependent drinkers and drug abusers. The brief motivational intervention will be tailored to the patient's age. Its purpose will be to motivate problem drinkers to change their drinking. The action-oriented moderation and abstinence protocols are cognitive-behavioral interventions (CBIs) that provide patients with the skills to maximize their chances of success with changing their drinking and/or drug use.

The investigators have already developed these elements but they are not integrated into a single program with appropriate branching between them. Nor has the content been tailored for use in primary care.

ELIGIBILITY:
Inclusion Criteria:

* physicians,
* nurses,
* nurse practitioners,
* physician's assistants,
* psychologists embedded in primary care settings, and
* other mental health counselors embedded in primary care settings.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Feasibility Questionnaire | Within 1 month of enrollment with an expected average of 1 week..
  A 17 item questionnaire that asks about the feasibility of using the web app with patients in primary care and the app's technical merit.

CONTACTS AND LOCATIONS:
Locations (1):
- Behavior Therapy Associates, LLC, Albuquerque, New Mexico, United States